CLINICAL TRIAL: NCT00708968
Title: Prostate Cancer: Family Care for Patients and Spouses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Laurel L. Northouse PhD/ Professor of Nursing, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01CA090739 (NIH); R01CA090739 (NIH); UMCC 0080; IRBMED 2001-0091
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2008-07

CONDITIONS: Prostate Cancer; Quality of Life; Cancer Survivorship
Keywords: randomized clinical trial; coping; quality of life; family; family caregiver; cancer survivorship; communication; uncertainty; support; family education; Caregivers
MeSH Terms: conditions — Prostatic Neoplasms; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOCUS Intervention (Experimental): Dyads randomized to this arm received the FOCUS Program, 3 home visits and 2 phone calls by trained nurses.
  Interventions: Behavioral: FOCUS Program
- Standard Care (No Intervention)

INTERVENTIONS:
Behavioral: FOCUS Program — Supportive, educative sessions with patients and spouses.
  Other Names: Prostate Cancer Patient and Spouse Intervention; Family-based intervention
  Arms: FOCUS Intervention

SUMMARY:
The purpose of this study is to determine if a family-based intervention (The FOCUS Program) can improve the long-term quality of life and other psycho-social outcomes of men with prostate cancer and their spouses.

DETAILED DESCRIPTION:
The purpose of this study was to determine if a family-based intervention (The FOCUS Program) could improve the long-term quality of life and other psycho-social outcomes of men with prostate cancer and their spouse/partners. Aim 1. The first aim was to determine if the family intervention could improve several proximal clinical outcomes (less negative appraisal of illness or caregiving, less uncertainty, less hopelessness, better family communication, higher self-efficacy, and more problem-focused coping) and improve the distal clinical outcome, quality of life, in a culturally and economically diverse sample of men with prostate cancer and their spouses. Aim 2. The second aim was to test a stress-coping model designed to predict which prostate cancer patients and their spouses are at higher risk of poorer long-term quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of prostate cancer
* Willing spousal partner
* Speaks and understands English
* Mentally and physically able to participate
* Minimum life expectancy of 12 months
* Lives within 70 miles

Exclusion Criteria:

* Multiple primary cancers
* Watchful waiting status
* Spouse with cancer diagnosis in previous year

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2001-09; Primary Completion 2005-10 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Baseline, 4, 8 and 12 months

SECONDARY OUTCOMES:
Threat appraisal | Baseline, 4, 8 and 12 months
Uncertainty | Baseline, 4, 8 and 12 months
Hopelessness | Baseline, 4, 8 and 12 months
Coping | Baseline, 4, 8 and 12 months
Family Communication | Baseline, 4, 8 and 12 months
Self-Efficacy | Baseline, 4, 8 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurel L Northouse, PhD RN, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University-Karmanos Cancer Institute, Detroit, Michigan
  - William Beaumont Hospitals, Royal Oak, Michigan

REFERENCES:
- [Background] Northouse LL, Rosset T, Phillips L, Mood D, Schafenacker A, Kershaw T. Research with families facing cancer: the challenges of accrual and retention. Res Nurs Health. 2006 Jun;29(3):199-211. doi: 10.1002/nur.20128. PMID 16676337
- [Background] Harden J, Falahee M, Bickes J, Schafenacker A, Walker J, Mood D, Northouse L. Factors associated with prostate cancer patients' and their spouses' satisfaction with a family-based intervention. Cancer Nurs. 2009 Nov-Dec;32(6):482-92. doi: 10.1097/NCC.0b013e3181b311e9. PMID 19816159
- [Background] Kershaw TS, Mood DW, Newth G, Ronis DL, Sanda MG, Vaishampayan U, Northouse LL. Longitudinal analysis of a model to predict quality of life in prostate cancer patients and their spouses. Ann Behav Med. 2008 Oct;36(2):117-28. doi: 10.1007/s12160-008-9058-3. Epub 2008 Sep 16. PMID 18830672
- [Background] Song L, Northouse LL, Braun TM, Zhang L, Cimprich B, Ronis DL, Mood DW. Assessing longitudinal quality of life in prostate cancer patients and their spouses: a multilevel modeling approach. Qual Life Res. 2011 Apr;20(3):371-81. doi: 10.1007/s11136-010-9753-y. Epub 2010 Oct 8. PMID 20927648
- [Background] Song L, Northouse LL, Zhang L, Braun TM, Cimprich B, Ronis DL, Mood DW. Study of dyadic communication in couples managing prostate cancer: a longitudinal perspective. Psychooncology. 2012 Jan;21(1):72-81. doi: 10.1002/pon.1861. Epub 2010 Oct 22. PMID 20967920
- [Result] Northouse LL, Mood DW, Schafenacker A, Montie JE, Sandler HM, Forman JD, Hussain M, Pienta KJ, Smith DC, Kershaw T. Randomized clinical trial of a family intervention for prostate cancer patients and their spouses. Cancer. 2007 Dec 15;110(12):2809-18. doi: 10.1002/cncr.23114. PMID 17999405
- [Result] Northouse LL, Mood DW, Montie JE, Sandler HM, Forman JD, Hussain M, Pienta KJ, Smith DC, Sanda MG, Kershaw T. Living with prostate cancer: patients' and spouses' psychosocial status and quality of life. J Clin Oncol. 2007 Sep 20;25(27):4171-7. doi: 10.1200/JCO.2006.09.6503. Epub 2007 Jul 16. PMID 17635953
- See also: University of Michigan Comprehensive Cancer Center website — http://www.cancer.med.umich.edu/